CLINICAL TRIAL: NCT04997226
Title: Cognitive Enhancement in Healthy Elderly People
Acronym: Pro-Cog
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bar-Ilan University, Israel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 04102020
Record Dates: First submitted 2021-08-02; First posted 2021-08-09 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-02

CONDITIONS: Transcranial Direct Current Stimulation; Transcranial Alternating Current Stimulation
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: The investigators will compare 4 intervention protocols aiming to improve memory performance:
  tDCS over the left DLPFC with adaptive memory game; Sham-tDCS with adaptive memory game; tACS over the left DLPFC at theta-gamma coupling with adaptive memory game; Sham tACS over the left DLPFC at theta-gamma coupling with adaptive memory game
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are randomly assigned to one of the four groups and are not aware whether they receive sham or real stimulation.
  Data analysis will be conducted with analysts blind to the study condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- tDCS over the left DLPFC with adaptive memory game (Active Comparator): The stimulation will be carried out using a battery-powered mobile device made by "Neurocon" with two 5 x 5 cm electrodes The anodal electrode will be positioned above the F3 region of a standard EEG cap that is parallel to the cortical DLPFC region. The return electrode will be placed over the right eyebrow. The electrodes will remain on the subjects head for 50 minutes - the entire duration of the session. 1mA stimulation will be given for 15 minutes, then a 20-minute break and again 15 minutes of 1 mA stimulation. This protocol has been shown to improve the duration of the stimulus effect (Monte-Silva et al., 2013).
  Interventions: Device: tDCS or tACS over the left DLPFC with adaptive memory game
- Sham tDCS over the left DLPFC with adaptive memory game (Placebo Comparator): As above but current will be operated for 1 minute - 30 seconds ramp up to 1 mA and 30 seconds ramp-down to initiate similar sensations to real stimulation. The electrodes will stay on the subjects heads for 50 minutes, similar to the active tDCS arm.
  Interventions: Device: Sham tDCS or tACS over the left DLPFC with adaptive memory game
- tACS over the left DLPFC at theta-gamma coupling with adaptive memory game (Active Comparator): As above but stimulation method will be employed at 2mA intensity for 20 minutes at theta-gamma coupling using a laplacian montage (Alekseichuk et al., 2016).
  Interventions: Device: tDCS or tACS over the left DLPFC with adaptive memory game
- Sham tACS over the left DLPFC at theta-gamma coupling with adaptive memory game (Placebo Comparator): As above but current will be operated for 1 minute - 30 seconds ramp up to 1 mA and 30 seconds ramp-down to initiate similar sensations to real stimulation. The electrodes will stay on the subjects heads for 20 minutes, similar to the active tACS arm.
  Interventions: Device: Sham tDCS or tACS over the left DLPFC with adaptive memory game

INTERVENTIONS:
Device: tDCS or tACS over the left DLPFC with adaptive memory game — This intervention is described in arms 1 and 3.
  Arms: tACS over the left DLPFC at theta-gamma coupling with adaptive memory game; tDCS over the left DLPFC with adaptive memory game
Device: Sham tDCS or tACS over the left DLPFC with adaptive memory game — This intervention is described in arms 2 and 4.
  Arms: Sham tACS over the left DLPFC at theta-gamma coupling with adaptive memory game; Sham tDCS over the left DLPFC with adaptive memory game

SUMMARY:
According to the European Commission Special Report, till 2030 it is expected ca. 40% increase of population aged 66-79. Increasing population of elderly people in modern society has suggested that more individuals are expected to suffer from cognitive deficits, as chronological aging is usually accompanied by declined cognition, in particular memory functions.

The cognitive decline reaches medical attention for about 5-25% of the elderly population (over 65 years of age) as they suffer from Mild Cognitive Impairment (MCI). MCI is usually referred to as an intermediate phase between the expected cognitive decline of normal aging and the pathological cognitive decline linked to dementia. In recent years, a new viewpoint argues that substantial improvement in cognitive function may be possible even in older age, using appropriately designed training programs. In the current project the investigators propose a potential intervention that might delay the onset of dementia by maintaining cognitive performance in general and improving in MCI in particular.

The current approach is to employ cognitive enhancement protocols, such as the combination of non-invasive, low intensity electrical stimulation and memory training aiming to preserve and ultimately improve cognitive abilities in MCI and healthy elderly.

DETAILED DESCRIPTION:
Aging is associated with several physiological changes that affect global functioning, daily activity and quality of life. For instance, cognitive functions progressively decline during normal aging, as evidenced by decreased episodic memory and working memory (WM) performance.

The above mentioned cognitive decline reaches medical attention for about 5-25% of the elderly population (over 65 years of age) as they suffer from Mild Cognitive Impairment (MCI). MCI is usually referred to as an intermediate phase between the expected cognitive decline of normal aging and the pathological cognitive decline linked to dementia. Around 46% of people with MCI develop dementia within three years, compared to 3% of the age-matched population. According to Peterson's initial definition (Petersen, 2004), The selected technique to improve cognition as the investigators propose here is transcranial non invasive brain stimulation (TES). The investigators will employ a couple of these techniques of neuromodulation that have proven to influence performance in different cognitive domains. Here the investigators propose to combine the investigators' expertise and to investigate the effects on cognition and health of brain stimulation-based treatment in MCI patients compared to matched healthy controls, combine it with cognitive training and explore the longer term effects of the intervention.

Objectives. The main objective of the proposed research is to explore the potential intervention based on non-invasive brain stimulation and cognitive training to improve cognition in the elderly. In particular the investigators aim to explore:

1. The immediate efficacy of various stimulation protocols with cognitive training on cognitive improvement in the elderly.
2. The long term effect of a selected stimulation protocol on MCI improvement in the elderly.

According to a large controlled study on cognitive stimulation for people with MCI, the treatment proved effective in improving the functioning in several cognitive areas compared to a control group (Ball et al., 2002).The cognitive training in this study included a computerized training, which is more enjoyable and effective than pencil-and paper training due to its immediate feedback and engaging nature. In their systematic review of 26 studies on computerized cognitive training (CCT) for older people with known MCI, Hill et al. (2016) concluded that CCT is an efficient tool for cognitive enhancement in older people with MCI. The overall effect size on cognition score was moderate (Hedges' g=0.35); a large significant effect size on working memory; and there were moderate significant effect sizes for specific cognitive domains, such as verbal memory, non-verbal learning, attention and on psychological functioning measures. In contrast, and consistent with findings of previous CCT meta-analysis (Motter, Pimontel et al., 2016), there were insignificant results regarding executive functions, processing speed and non-verbal memory. The results on dementia patients, as opposed to MCI ones, were less optimistic: there was only a small but statistically significant effect size of the overall efficacy of the CCT on cognition enhancement.

The researchers have previous works that revealed an enhanced training effect when it was combined with non-invasive brain stimulation, for example better cognitive control following training combined with Transcranial direct current stimulation (tDCS) compared to training alone (Ditye et al., 2012).

Transcranial direct current stimulation (tDCS) is a safe, low-cost, non-invasive neurophysiological technique that consists in the application of mild (1-2 milliampere (mA)) electrical current on the scalp (Jacobson et al., 2012).

There is growing evidence that tDCS, combined with cognitive stimulation, improves cognitive functioning among healthy adult subjects. Specifically, tDCS to the prefrontal cortex has been proved effective. Anodal stimulation of the left dorsolateral prefrontal cortex (DLPFC) increases the performance on a working memory task in young healthy adults. In a combined treatment of behavioral training and tDCS stimulation of ten sessions for 10 days, healthy elderly subjects increased working memory skills for up to 28 days (Park et al., 2014).

tDCS has also been proved efficient for people with Alzheimer's Disease (AD) or other types of dementia. In one study, anodal tDCS was applied to both hemispheres of the temporal cortex in 30 minutes sessions for five successive days. Results showed a significant improvement in a visual recognition memory task. tDCS anodal stimulation of the Broca's region within the left inferiorfrontal gyrus (IFG) had some positive effects on verbal fluency among patients with MCI in a double-blind, crossover, sham-controlled stimulation study. Additional brain imaging analysis of these results indicated that there was also a reduction of compensatory upregulated activity within the frontal cortices. Manenti et al. (2016) have used anodal tDCS combined with physical therapies in MCI patients with Parkinson's disease (PD). Following daily administration of 2 mA stimulation for two weeks, subjects have improved their PD Cognitive Rating Scale scores and their verbal fluency test, in comparison with the sham control group.

The efficacy of using tDCS in combination with cognitive training is yet controversial. A study on AD patients which used anodal tDCS to stimulate the left DLPFC in a name-face association learning task, found no additional effect to the tDCS stimulation beyond that of the behavioral training. In contrast to these findings, in a study of healthy subjects, the combination of tDCS stimulation and simultaneous cognitive behavioral training has been proved more effective than tDCS stimulation to the left DLPFC by itself (Martin, Liu, Alonzo et al., 2015).

In a recent study (André et al., 2016), four sessions of anodal tDCS stimulation over the left DLPFC, in combination with different cognitive tasks, were applied to 21 patients with mild vascular dementia. There was a significant improvement up to two weeks later in visual short term memory (in a pictures naming task), verbal working memory (2-back task) and executive control (go/no go task) in the anodal stimulation group, Yet, there are still some considerable limitations to the research on tDCS effects on cognition and to its clinical applications. For instance, choosing the target area or network is, of course, critical. Various target areas have been used in different studies: frontal lobe, especially the DLPFC and the IFG, are natural candidates. Few studies have targeted the inferior parietal lobe, which might require further research.

To overcome some of the problems the investigators will test another brain stimulation technique, transcranial alternating current stimulation (tACS) where promising previous results suggest that tACS over prefrontal areas might be a better tool to improve cognitive functions in the elderly. tACS, a specific subtype of Non-invasive Brain Stimulation methods (NIBS), is based on the application of low-intensity electrical currents oscillating sinusoidally at a predetermined frequency (Antal et al., 2008). TACS-mediated physiological and behavioral changes seems to be frequency-dependent, thus, tACS could interact with the on-going brain activity through cortical oscillatory entrainment.

Since episodic memory decline is one of the most important markers of MCI, the investigators will test brain stimulation protocols that were found to affect different types of memory performance. Possible effects of transcranially applied oscillating currents on memory functions have been investigated on humans by using transcranial Slow Oscillation Stimulation (SO-tDCS; i.e., anodal transcranial direct current stimulation oscillating at 0.75 Hz in a trapezoid waveform-fashion, applied bi-frontally) in combination with on-line EEG recording during slow wave sleep (Marshall et al., 2006). Ripple-range oscillations in the hippocampus have also been associated with declarative memory consolidation. The co-PI, Prof. Antal reported that bilateral 140 Hz tACS over both DLPFC during encoding may have a positive effect on the consolidation of declarative material (Ambrus et al., 2015). Novel cross-frequency protocols (theta-gamma coupling) of tACS affected spatial working memory performance in humans: enhancement of working memory performance and increase of global neocortical connectivity were observed when bursts of high gamma oscillations (80-100 Hz) coincided with the peaks of the theta waves, whereas superimposition on the trough of the theta wave and low gamma frequency protocols were ineffective.

In sum, evidence from recent studies portray a promising picture of this new line of research, suggesting that non-invasive brain stimulation techniques, in general, and tDCS and tACS, in particular, may be used to ameliorate cognitive dysfunction in patients in pre-dementia. Though prospects seem promising, the mixed results and inconclusive findings of several studies call for cautious. Hopefully, the proposed research will narrow the gap between theoretical knowledge and the clinical applicability of the findings for the sake of a treatment that can truly affect many people's lives.

The current approach is to employ cognitive enhancement tools aiming to develop effective protocols that will preserve (and ultimately improve) cognitive abilities in MCI and healthy elderly. The main method are non-invasive brain stimulation tools, tDCS and tACS, combined with computer-based cognitive training in a multiple session design.

Patient Registries:

Each subject is met by the experimenters (PhD students) for 16 individual meetings. The baseline measurements and cognitive evaluation that is manually conducted by the experimenters is inserted and saved in local Excel files. The subjects' performance in the computerized games (the cognitive training) is automatically saved on the lab's computer.

Quality assurance: the completeness and accuracy of the training log files is checked after every session.

Standard Operating Procedures - a paper file is prepared for each subject to keep background and contact details, printed records of the subjects' performance in the memory evaluation tests (at baseline, immediately after completing the intervention, and 3 months after completing the intervention).

Sample size assessment: The sample size was a priori calculated using More Power software (Campbell & Thompson, 2012) based on the effect size reported for memory enhancement by transcranial electrical stimulation by Jacobson et al. (2012) (d = 0.49). This established that with a α = 0.05, power = 0.95, 60 participants are necessary to detect a moderate-large effect.

Statistical analysis plan: data will be analyzed with IBM Statistical Package for Windows, version 23 (IBM Corp., Armonk, N.Y., USA). The main analysis is a mixed design analysis that compares the experimental conditions (between subject factors) regarding their effect on memory performance in 2 episodic memory tests and 3 time points (within subjects variables). The cognitive status at baseline will serve as a covariate (the baseline scores). In addition, the investigators plan hierarchical regression to check how ongoing scores in the cognitive training predict episodic memory score at the end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

normal or corrected-to-normal vision good general health independent living MoCa score of at least 24 -

Exclusion Criteria:

A history of acute or chronic neurological illness, heart disease, metabolic disorders, vascular disorders psychiatric disorder. epilepsy metal implants

-

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Visual episodic memory of word pairs learning test (Marshall et al., 2004) | Change from baseline (before treatment) to immediately after treatment (6 weeks) and 3 months after end of treatment
  Number of correctly recalled word pairs
Ray auditory verbal learning test (episodic memory) includes immediate recall, and after time (Carlesimo et al., 1996), | Change from baseline (before treatment) to immediately after treatment (6 weeks) and 3 months after end of treatment
  Number of correctly recalled items

SECONDARY OUTCOMES:
Logical Memory Test 1 (Craft et al., 2000; Wechsler, 2008) | Change from baseline (before treatment) to immediately after treatment (6 weeks) and 3 months after end of treatment
  Number of correctly recalled items
Montreal questionnaire for Cognitive Assessment (MoCA, Nasreddine et al., 2005) | Change from baseline (before treatment) to immediately after treatment (6 weeks) and 3 months after end of treatment
  Score at the MoCA test

CONTACTS AND LOCATIONS:
Overall Officials: Michal Lavidor, Prof., Principal Investigator — Bar Ilan University
Locations (1):
- Department of Psychology, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No
The investigators will generate big data files due to 16 meetings with all 120 participants. There is not much point in sharing these mega-files, rather the investigators can share the final groups averages to measure memory change in the 4 experimental group

REFERENCES:
- [Result] Meiron O, Lavidor M. Prefrontal oscillatory stimulation modulates access to cognitive control references in retrospective metacognitive commentary. Clin Neurophysiol. 2014 Jan;125(1):77-82. doi: 10.1016/j.clinph.2013.06.013. Epub 2013 Jul 3. PMID 23831184
- [Result] Monte-Silva K, Kuo MF, Hessenthaler S, Fresnoza S, Liebetanz D, Paulus W, Nitsche MA. Induction of late LTP-like plasticity in the human motor cortex by repeated non-invasive brain stimulation. Brain Stimul. 2013 May;6(3):424-32. doi: 10.1016/j.brs.2012.04.011. Epub 2012 Jun 2. PMID 22695026
- [Result] Jacoby N, Lavidor M. Null tDCS Effects in a Sustained Attention Task: The Modulating Role of Learning. Front Psychol. 2018 Apr 6;9:476. doi: 10.3389/fpsyg.2018.00476. eCollection 2018. PMID 29681876
- [Result] Jacobson L, Koslowsky M, Lavidor M. tDCS polarity effects in motor and cognitive domains: a meta-analytical review. Exp Brain Res. 2012 Jan;216(1):1-10. doi: 10.1007/s00221-011-2891-9. Epub 2011 Oct 12. PMID 21989847
- [Result] Ditye T, Jacobson L, Walsh V, Lavidor M. Modulating behavioral inhibition by tDCS combined with cognitive training. Exp Brain Res. 2012 Jun;219(3):363-8. doi: 10.1007/s00221-012-3098-4. Epub 2012 Apr 25. PMID 22532165
- [Result] Petersen RC. Mild cognitive impairment as a diagnostic entity. J Intern Med. 2004 Sep;256(3):183-94. doi: 10.1111/j.1365-2796.2004.01388.x. PMID 15324362
- [Result] Ball K, Berch DB, Helmers KF, Jobe JB, Leveck MD, Marsiske M, Morris JN, Rebok GW, Smith DM, Tennstedt SL, Unverzagt FW, Willis SL; Advanced Cognitive Training for Independent and Vital Elderly Study Group. Effects of cognitive training interventions with older adults: a randomized controlled trial. JAMA. 2002 Nov 13;288(18):2271-81. doi: 10.1001/jama.288.18.2271. PMID 12425704
- [Result] Hill NT, Mowszowski L, Naismith SL, Chadwick VL, Valenzuela M, Lampit A. Computerized Cognitive Training in Older Adults With Mild Cognitive Impairment or Dementia: A Systematic Review and Meta-Analysis. Am J Psychiatry. 2017 Apr 1;174(4):329-340. doi: 10.1176/appi.ajp.2016.16030360. Epub 2016 Nov 14. PMID 27838936
- [Result] Motter JN, Pimontel MA, Rindskopf D, Devanand DP, Doraiswamy PM, Sneed JR. Computerized cognitive training and functional recovery in major depressive disorder: A meta-analysis. J Affect Disord. 2016 Jan 1;189:184-91. doi: 10.1016/j.jad.2015.09.022. Epub 2015 Sep 26. PMID 26437233
- [Result] Park SH, Seo JH, Kim YH, Ko MH. Long-term effects of transcranial direct current stimulation combined with computer-assisted cognitive training in healthy older adults. Neuroreport. 2014 Jan 22;25(2):122-6. doi: 10.1097/WNR.0000000000000080. PMID 24176927
- [Result] Manenti R, Sandrini M, Brambilla M, Cotelli M. The optimal timing of stimulation to induce long-lasting positive effects on episodic memory in physiological aging. Behav Brain Res. 2016 Sep 15;311:81-86. doi: 10.1016/j.bbr.2016.05.028. Epub 2016 May 13. PMID 27185737
- [Result] Martin DM, Liu R, Alonzo A, Green M, Loo CK. Use of transcranial direct current stimulation (tDCS) to enhance cognitive training: effect of timing of stimulation. Exp Brain Res. 2014 Oct;232(10):3345-51. doi: 10.1007/s00221-014-4022-x. Epub 2014 Jul 4. PMID 24992897
- [Result] Andre S, Heinrich S, Kayser F, Menzler K, Kesselring J, Khader PH, Lefaucheur JP, Mylius V. At-home tDCS of the left dorsolateral prefrontal cortex improves visual short-term memory in mild vascular dementia. J Neurol Sci. 2016 Oct 15;369:185-190. doi: 10.1016/j.jns.2016.07.065. Epub 2016 Jul 30. PMID 27653887
- [Result] Antal A, Boros K, Poreisz C, Chaieb L, Terney D, Paulus W. Comparatively weak after-effects of transcranial alternating current stimulation (tACS) on cortical excitability in humans. Brain Stimul. 2008 Apr;1(2):97-105. doi: 10.1016/j.brs.2007.10.001. Epub 2007 Dec 3. PMID 20633376
- [Result] Marshall L, Helgadottir H, Molle M, Born J. Boosting slow oscillations during sleep potentiates memory. Nature. 2006 Nov 30;444(7119):610-3. doi: 10.1038/nature05278. Epub 2006 Nov 5. PMID 17086200
- [Result] Ambrus GG, Pisoni A, Primassin A, Turi Z, Paulus W, Antal A. Bi-frontal transcranial alternating current stimulation in the ripple range reduced overnight forgetting. Front Cell Neurosci. 2015 Sep 24;9:374. doi: 10.3389/fncel.2015.00374. eCollection 2015. PMID 26441544
- [Result] Campbell JI, Thompson VA. MorePower 6.0 for ANOVA with relational confidence intervals and Bayesian analysis. Behav Res Methods. 2012 Dec;44(4):1255-65. doi: 10.3758/s13428-012-0186-0. PMID 22437511
- [Derived] Ben Izhak S, Jacoby N, Diedrich L, Antal A, Lavidor M. Enhanced cognitive performance in older adults through combined cognitive training and transcranial direct current stimulation. Sci Rep. 2025 Jul 6;15(1):24114. doi: 10.1038/s41598-025-08322-6. PMID 40619473